CLINICAL TRIAL: NCT06259708
Title: Effectiveness of Targeting the Zona Incerta (ZI) for Tremor Control in Parkinson's Disease Patients
Brief Title: Using Low Intensity Focused Ultrasound to Modulate Deep Brain Areas for Tremor Control in Parkinson's Disease Patients.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Focused Ultrasound Foundation (Other)
Responsible Party: Principal Investigator, Martin McKeown, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: H23-00480
Record Dates: First submitted 2024-01-26; First posted 2024-02-14 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
Keywords: Low intensity focused ultrasound; Parkinsons disease; Tremor; Zona incerta
MeSH Terms: conditions — Parkinson Disease; Tremor

STUDY DESIGN:
Intervention Model Description: The investigators will use a crossover design for this study as it requires fewer participants and removes variance between participants in the outcomes that are irrelevant to the stimulation type in comparison to other designs where each participant only receives one stimulation. All participants receive all the stimulation types (Vim-LIFU and ZI-LIFU), but the order in which they get the stimulation types is randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vim first (Experimental): Participants assigned to this arm get LIFU stimulation in the Vim before the ZI.
  Interventions: Device: Low intensity focused ultrasound
- ZI first (Experimental): Participants assigned to this arm get LIFU stimulation in the Vim before the ZI.
  Interventions: Device: Low intensity focused ultrasound

INTERVENTIONS:
Device: Low intensity focused ultrasound — Sonication with low intensity focused ultrasound in two deep brain structures (ZI and Vim).

SUMMARY:
Researchers have found that a treatment called Magnetic Resonance guided Focused Ultrasound (MRgFUS) can effectively reduce tremors in patients with essential tremor (ET) and Parkinson's disease (PD). They noticed that ET patients initially responded better to the treatment than PD patients, but by the end of the treatment, both groups showed similar improvement. The study also suggested that targeting a specific area of the brain called the Zona Incerta (ZI) may be more beneficial for PD patients. Based on these findings, the investigators plan to use low-intensity focused ultrasound to directly modulate the ZI area and investigate the mechanisms of reduced tremors in PD patients. The investigators will also compare the effectiveness of this approach with the current target, the ventral intermediate nucleus (Vim) of the thalamus. The investigators will use a simulation model to determine the best ultrasound parameters for this new approach and will also examine the impact of the treatment on the brain's network activity using functional Magnetic Resonance Imaging. Success of this project may lay the foundation for finding a more effective target for MRgFUS treatment of PD tremor.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Parkinson's disease
* Resting tremor score (MDS-UPDRS III 3.17 Rest Tremore Amplitude (RUE or LUE)) ≥ 2
* Between the ages of 40-80 years
* Hoehn and Yahr stage between 1-3 (mild to moderate PD) in the "ON" state
* Patients who are willing to have a partial (~8 cm diameter circular area above the ear) hair shaving.

Exclusion Criteria:

* Atypical Parkinsonism
* History of essential tremor
* Dementia preventing informed consent
* Change in Parkinson's medication with the last 2 weeks
* Neurological disease other than PD, including Alzheimer's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, a brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma
* Unstable medical conditions or serious disease/conditions (e.g., cancer undergoing active treatment, poorly controlled diabetes)
* Concurrent treatment for PD with Duodopa
* Concurrent treatment for PD with deep brain stimulation (DBS)
* Thickness of the temporal bone < 7 mm
* Individuals should also not participate if they have any of the following contraindications for undergoing fMRI scanning:
* Cardiac pacemaker, wires, or defibrillator
* Metal in eye or orbit, including the history of any eye injury involving metal fragments and increased risk due to (history of) working as a metal worker (grinding, machining, or welding)
* Ferromagnetic aneurysm clip
* Possibility of pregnancy
* Artificial heart valve
* Ear or eye implant, including cochlear implant
* Brain aneurysm clip
* Implanted drug infusion pump
* Electrical stimulator to nerves or bones
* Coil, catheter, or filter in any blood vessel
* Orthopedic hardware (artificial joint, plate, screw, rod)
* Other metallic prostheses
* Shrapnel, bullets, or other metal fragments
* Surgery, piercings or tattoos (including tattooed eyeliner) in the last six weeks
* Medication releasing skin patches (i.e. nicotine, birth control, nitroglycerine)
* History of claustrophobia

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Tremor | At 50Hz for 40 minutes 30 minutes after intervention
  Finger displacement (angle [deg]).
Tremor | At 50Hz for 40 minutes 30 minutes after intervention
  Finger acceleration (mm/s^2)
Functional connectivity | Once before and once immediately after intervention
  fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Hongchae Baek, PhD, Principal Investigator — Food and Drugs Administration; Soojin Lee, PhD, Principal Investigator — University of British Columbia; Martin J. McKeown, MD, FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, DMCBH, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No